CLINICAL TRIAL: NCT04245150
Title: Assessing the Impact of the Microbiome on Breast Cancer Radiotherapy Toxicity
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE5118
Record Dates: First submitted 2019-12-20; First posted 2020-01-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: DCIS; Invasive Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast skin and GI samples from participants with breast cancer following breast conserving surgery will be collected. These samples will then be analyzed using DNA extraction and 16S rRNA gene sequencing with an in-house bioinformatics group. Data will be used to define the microbiome profile for this subset of breast cancer patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ductal Carcinoma In Situ (DCIS) or invasive breast cancer: Participants with DCIS or invasive breast cancer
  Interventions: Other: Stool sample; Other: Skin Swab Sample

INTERVENTIONS:
Other: Stool sample — Stool sample
Other: Skin Swab Sample — Skin Swab Sample

SUMMARY:
Microorganisms in the human body (such as virus, bacteria, fungus) may have an important role in breast cancer side effects. In this study, microorganisms will be analyzed to determine which, if any,are present. It will then be determined if side effects from breast radiation are associated with these microorganisms. Understanding the association of microorganisms with side effects will allow the study team to look at strategies to reduce side effects for patients undergoing radiation to the breast.

DETAILED DESCRIPTION:
This study will prospectively enroll 50 participants with with biopsy proven Ductal carcinoma in situ (DCIS) or invasive breast cancer 18 years of age or older, undergoing breast conserving surgery and adjuvant radiation therapy at Cleveland Clinic.

Each participant will have a post-surgery pre-radiotherapy stool and breast skin sample obtained, complete a medical record review for clinical data, and have complete an interview/questionnaire in order to learn about potential risk factors which will be included in the data collection form. Included information will include Stage (T, N, M, composite), receipt of chemotherapy, radiation fields and dose, BMI, hypertension (HTN), Diabetes Mellitus (DM), smoking status, history of breast infection yes/no (Data Collection Form).

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients with DCIS or invasive breast cancer
* Undergoing breast conserving surgery and adjuvant radiation
* Subjects must be willing and able to provide breast skin samples

Exclusion Criteria:

* Active clinical breast infection (on antiobiotic for skin/breast infection or clinical diagnosis)
* Refuse or are unable to sign informed consent form
* Past history of breast cancer

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy proven DCIS or invasive breast cancer, 18 years of age or older, undergoing breast conserving surgery and adjuvant radiation therapy at Cleveland Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Microbiome profile as assessed by stool sample | At baseline
  Microbiome profile as assessed by stool sample. Sample analysis will be done via DNA extraction and rRNA gene sequencing of stool sample
Microbiome profile as assessed by breast skin sample | At baseline
  Microbiome profile as assessed by breast skin sample. Sample analysis will be done via DNA extraction and rRNA gene sequencing of stool sample
Correlation of the microbiome to incidence of at least grade 3 skin toxicity using the CTCAE version 4.0 scoring | 3 months post-treatment
  The microbiome profiles identified will be correlated with incidence of at least grade 3 skin toxicity using the CTCAE version 4.0 scoring by visual assessment. Maximum toxicity during radiation will be recorded.
  Grade 0: None Grade 1: Faint erythema or dry desquamation Grade 2: Moderate to brisk erythema; patchy moist desquamation, mostly confined to skin folds and creases; moderate edema Grade 3: Moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion Grade 4: Life-threatening consequences; skin necrosis or ulceration of full thickness dermis; spontaneous bleeding from involved site; skin graft indicated

CONTACTS AND LOCATIONS:
Overall Officials: Chirag Shah, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States